CLINICAL TRIAL: NCT01882010
Title: Leukine (Sargramostim) for Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Sanofi (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Nebraska Neuroscience Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0487-12-FB; 2R01NS034239 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; motor function; immune activation; T cells; CD4; GMCSF; leukine; sargramostim; magnetoencephalography
MeSH Terms: conditions — Parkinson Disease | interventions — sargramostim; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Controls (Sham Comparator): Caregivers, spouse, friends, relatives of PD patients, have blood draws, MEG.
  Interventions: Diagnostic Test: Sham Comparator: Controls
- PD Patients placebo (Placebo Comparator): PD patients that receive placebo, have blood draw, physical exam and UPDRS part III assessment, MEG, Motion analysis.
  Interventions: Drug: placebo
- PD Patients sargramostim (Experimental): PD patients that receive Leukine, have blood draw, physical exam and UPDRS part III assessment, MEG, Motion analysis.
  Interventions: Drug: sargramostim

INTERVENTIONS:
Drug: sargramostim — lyophilized 250 micrograms/vial
  6 micrograms/kg daily subcutaneous injection
  56 days
  Other Names: Leukine
  Arms: PD Patients sargramostim
Drug: placebo — saline solution daily subcutaneous injection 56 days
  Other Names: saline solution
  Arms: PD Patients placebo
Diagnostic Test: Sham Comparator: Controls — Caregivers, spouse, friends, relatives of PD patients, have blood draws, MEG.
  Arms: Controls

SUMMARY:
The purpose of this study is to determine if Leukine (sargramostim) can be safely administered to Parkinson's disease patients for an extended period of time (56 days) and restore immune deficits seen in Parkinson's patients compared to controls. The development of magnetoencephalography (MEG) as a monitoring tool for PD will also be explored. At enrollment and repeating again at two 4-week intervals, whole blood from PD patients and controls will be obtained for analyses and the results will be used to calculate immune response profiles as a baseline for comparison after drug treatment. Physical examinations and motor assessments will also be performed on PD patients. After the 8-week baseline data collection, control participation will end and drug treatment of PD patients will begin. PD patients will be randomized, and half will receive drug and half will receive placebo. Leukine at a dosage of 6 µg/kg or saline as placebo will be administered by subcutaneous injection daily for 56 days (8 weeks). During drug treatment, PD patients will be monitored every two weeks by physical examinations, motor assessments, and blood analyses. As follow-up, four weeks after drug administration has stopped, subjects will again have physical examinations, motor assessments, and blood analyses. MEG will be performed on PD patients and controls at the start of drug treatment, and on PD patients at the end of the drug treatment period and 4 weeks after drug is stopped. In addtion, at the second cohort of 8 PD subjects, we will evaluate the potential Leukine-induced motor control and mobility improvements. Also, levels of the neurotransmitters glutamate, glutamine, serotonin, acetylcholine, GABA, norepinephrine and epinephrine in serum/plasma will be analyzed to correlate with changes in motor function and drug treatment.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive and disabling neurological disorder involving the nigrostriatum and for which no cure is known. Evidence suggests that inflammation contributes, significantly, to the cause and/or progression of the disease. Studies in postmortem human brain, animal models, and human peripheral blood support the idea that the frequency and function of particular circulating T cell subsets are abnormal and worsen as disease progresses. This abnormality is linked specifically to increases in numbers of T effector neurodestructive cells (Teff) and to dysfunction of regulatory T cells (Treg) that control Teff. This imbalance tips the homeostatic balance to a pro-inflammatory profile with limited control. Nonetheless, whether such T cell deficits are a cause of PD or a reaction to it remains unknown. If these deficits are causal or exacerbative, then correcting the deficit could have significant positive effects on disease progression and could ameliorate nigrostriatal degeneration or its sequelae. Granulocyte macrophage colony stimulating factor (GM-CSF) is a potential immunomodulatory therapeutic for PD to increase Treg numbers or function and reduce or transform proinflammatory Teff responses, leading to neuroprotection of the nigrostriatum and improved clinical outcomes for disease. Recombinant human GM-CSF (sargramostim) is available as Leukine®. The purpose of this study is to determine if Leukine (sargramostim) can be safely administered to Parkinson's disease patients for an extended period of time (56 days).

In a previous study conducted at the University of Nebraska Medical Center (UNMC) using samples of whole blood, PD patients showed differences from caregiver controls according to results from complete blood count (CBC) with white blood cell (WBC) differential, fluorescence-activated cell sorting (FACS) analysis for T cell markers, and Treg functional assays. These immune aberrations correlated with motor dysfunction as determined by Parkinson's disease rating scale (UPDRS) part III assessments. In this pilot study, the effect of Leukine treatment on immune deficits in PD patients will be monitored. Immune cell analyses of whole blood, motor assessments, and physical examinations and blood analyses for safety, will be conducted before, during, and after Leukine or placebo treatment of PD patients, and using healthy controls during baseline data collection before drug treatment. Initially, 16 PD patients and 16 controls will be recruited. Subjects will be drawn from the previous study. Enrollment will be supplemented as needed with patients from Neurology Consultants of Nebraska-PC, UNMC Neurological Sciences, or recruitment through the American Parkinson's Disease Association. Enrollment will be staggered, and additional subjects will be recruited as needed to replace any withdrawing participants, with the goal of 32 subjects, 16 PD patients and 16 controls, completing the study.

At enrollment and repeating again at two 4-week intervals, whole blood from PD patients and controls will be obtained percutaneously using standard sterile techniques. CBC with WBC differential, FACS analysis for T cell markers, and Treg functional assays will be performed and used to calculate immune response profiles as a baseline for comparison after drug treatment. Blood chemistries will be analyzed including liver enzymes, electrolytes, blood urea nitrogen, creatinine, total protein, albumin and bilirubin levels, and anti-GM-CSF antibodies will be assessed in PD patients. PD patients will be evaluated by physical and clinical examinations, including UPDRS part III assessments for evaluation of motor function.

PD patients will then be randomized into two groups, placebo (n=8) and Leukine (n=8), and participation of the controls will end. Patients entered into the study will not have any noted co-morbid conditions including infection, inflammatory or cancerous diseases and will not be taking immunostimulatory or immunosuppressive medicines. Patients will continue to take medicines prescribed for the general treatment of PD, including, but not limited to, dopamine or dopamine agonists. There will be no history of prior surgeries linked to PD treatment. Patients will receive training for self-injection, and the treatment group will self-administer Leukine (6 µg/kg) by subcutaneous injection daily for eight weeks. The placebo group will self-administer saline as placebo. Every two weeks after the start of treatment and again 4 weeks after cessation of administration, all PD patients, receiving drug or placebo, will be evaluated by physical and clinical examinations, including UPDRS part III assessments. Every 2 weeks during Leukine treatment and again 4 weeks after cessation of drug, whole blood from PD patients will be obtained percutaneously using standard sterile techniques. At weeks 2, 4 and 8, results from CBC with WBC differential, FACS analysis for T cell markers, and Treg functional assays will be used to calculate immune response profiles and compared with baseline values. CBC with WBC differential, total T cell count, and blood chemistries will be analyzed every 2 weeks for evidence of potential toxicities, as well as 4 weeks after termination of Leukine treatment. Levels of anti-GM-CSF antibodies will be assessed for PD patients at enrollment and at 4 weeks intervals during drug treatment and 4 weeks after termination. Optional video recordings will be made at baseline, end of drug/placebo treatment and at follow-up.

An additional component of the study includes the development of magnetoencephalography (MEG) as a monitoring tool for PD. MEG provides a non-invasive method to study brain activity. Currently, there are not adequate assessment tools for monitoring disease progression or treatment protocols in PD. In preliminary experiments on PD patients and their caregivers, MEG data have indicated strong beta synchronization during rest in PD and milder beta desynchronization during movement preparation compared to age- and sex-matched controls. In this study, the amplitude of this pathological beta synchronization/desynchronization will be monitored to evaluate improvements in cortical brain function of PD patients treated with Leukine. MEG will be performed on PD patients and controls at the start of drug treatment, and on PD patients at the end of the drug treatment period and 4 weeks after drug is stopped.

Among the first 8 patients enrolled in the study, we have observed unexpected and statistically significant changes in the unified PD rating scale part III (UPDRS part III) clinical evaluations for motor function in half of the patients tested. This test, however, is viewed as subjective. To more objectively and analytically score motor functions, biomechanical assessments of the subject's mobility, postural balance, upper extremity motor control and resting state tremor will be performed on the remaining eight PD patients receiving Leukine or placebo. These assessments will occur at baseline, between 7 and 8 weeks of drug treatment, and at 4-5 weeks after cessation of drug treatment. Motor function tests are designed to provide an objective, computer generated score as measured by patient performance on each test. To investigate a possible mechanism for changes in motor function observed within two weeks of therapy, testing for plasma/serum neurotransmitters will be performed to include glutamate, glutamine, serotonin, acetylcholine, gamma-aminobutyric acid (GABA), norepinephrine and epinephrine. These measures will be performed on the last cohort of PD patients of the study before initiation of treatment, 8 weeks after treatment is initiated and at 4 weeks after cessation of drug treatment. The tests will be evaluated by enzyme-linked immunosorbent assay (ELISA) or by ultra-performance liquid chromatography (UPLC). A decision on which assay will be done for which neurotransmitter will be based on sensitivity and standard curve measures. Relationships between neurotransmitter levels and motor function will be determined. These tests are in addition to current ongoing and approved laboratory tests. Eligibility requirements are unchanged from those currently imposed. Measures of motor function and serum/plasma neurotransmitter concentrations will also be completed 4-5 weeks after cessation of treatment. The notion of exploring neurotransmitters in this study is based on role in motor function that include fatigue, bowel, sexual dysfunction and mood changes that are also observed in PD as well as that GM-CSF has been shown to affect neurotransmitter levels (96). This range of listed neurotransmitters was not investigated in the first part of this study and will require limited additional blood and assay resources for the last part of the investigation.

ELIGIBILITY:
Inclusion Criteria:

PD Patients

* Onset of bradykinesia and 1 or both of the following: rest tremor and/or rigidity
* Asymmetric onset of clinical signs
* Progressive motor symptoms
* Age at onset 35-85 years
* Duration of PD symptoms of at least 3 years
* Female subjects must be either:

Not pregnant, not breastfeeding, and not planning on becoming pregnant during the study; Not of childbearing potential, defined as one who has been postmenopausal for at least 1 year and with follicle stimulating hormone (FSH) levels in the laboratory defined postmenopausal range, or has been surgically sterilized, or has had a hysterectomy at least 3 months prior to the start of this trial; or If of childbearing potential, must agree to use an effective method of avoiding pregnancy to the end of the trial and must have a negative serum beta-human chorionic gonadotropin (β-HCG) test. Effective methods of avoiding pregnancy are contraceptive methods used consistently and correctly (including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragm with spermicide, male or female condoms with spermicide, or cervical cap), abstinence, or a sterile sexual partner

* Have the ability to comply with basic instructions and have the ability to sit still comfortably inside the MEG
* Must be stage 4 or less according to the Hoehn and Yahr scale
* Caregiver, spouse, friend, or relative must agree to participate in the research study

Control subjects:

* Age 35-85 years
* Caregiver, spouse, relative, or friend of eligible PD patient
* Female subjects must be either:

Not pregnant, not breastfeeding, and not planning on becoming pregnant during the study; Not of childbearing potential, defined as one who has been postmenopausal for at least 1 year and with follicle stimulating hormone (FSH) levels in the laboratory defined postmenopausal range, or has been surgically sterilized, or has had a hysterectomy at least 3 months prior to the start of this trial; or If of childbearing potential, must agree to use an effective method of avoiding pregnancy to the end of the trial and must have a negative serum beta-human chorionic gonadotropin (β-HCG) test. Effective methods of avoiding pregnancy are contraceptive methods used consistently and correctly (including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragm with spermicide, male or female condoms with spermicide, or cervical cap), abstinence, or a sterile sexual partner

* Have the ability to comply with basic instructions and have the ability to sit still comfortably inside the MEG

Exclusion Criteria:

PD Patients

* Atypical features indicative of a Parkinson-Plus disorder (Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD)) including cerebellar signs, supranuclear gaze palsy, apraxia and other cortical signs, or prominent autonomic failure
* Neuroleptic treatment at time of onset of parkinsonism
* Active treatment with a neuroleptic at time of study entry
* History of repeated strokes with stepwise progression of parkinsonism
* History of repeated head injury
* History of definite encephalitis
* More than one blood relative diagnosed with PD
* Prominent gait imbalance early in the course (< 5 years)
* Mini-mental state examination score <26
* Hematological malignancy or coagulopathy
* Abnormal blood analyses: hematocrit <30; WBC>11.5; clinically significant laboratory data (e.g. alanine aminotransferase [ALT] or aspartate aminotransferase [AST] 3x the upper limit of normal [ULN]), or any abnormal laboratory value that could interfere with the assessment of safety in the judgment of the investigator; significant abnormalities on the clinical examination, vital signs, and clinical chemistry or hematology results (excluding findings of Parkinson's disease), that may interfere with the study or present a safety risk for the subject as judged by the clinical investigator charged in the care of study participants
* Serious medical illness or co-morbidity that may interfere with participation in the study
* Brain surgery for parkinsonism (DBS, cell implantation, gene therapy)
* History of an autoimmune disorder or systemic inflammatory disorder
* Immunostimulatory or immunosuppressive treatment (including amphetamines or systemic corticosteroids) within 90 days
* Exclusively unilateral parkinsonism for longer than 3 years
* Known hypersensitivity to GM-CSF, yeast-derived products or benzyl alcohol
* Current lithium treatment
* Individuals who have ferrous metal implanted in their body other than fillings
* Individuals with current diagnoses of alcohol or substance abuse/dependence
* Anyone who is not appropriate for participation in this research protocol as deemed by the principal or co-investigator

Control subjects:

* Positive response to more than 3 items on the PD Screening Questionnaire
* More than one blood relative diagnosed with by PD
* Mini-mental state examination score <26
* Hematological malignancy or coagulopathy
* Abnormal blood analyses: hematocrit <30; WBC>11.5; clinically significant laboratory data (e.g. alanine aminotransferase [ALT] or aspartate aminotransferase [AST] 3x the upper limit of normal [ULN]), or any abnormal laboratory value that could interfere with the assessment of safety in the judgment of the investigator; significant abnormalities on the clinical examination, vital signs, and clinical chemistry or hematology results that may interfere with the study or present a safety risk for the subject as judged by the investigator
* Serious medical illness or comorbidity that may interfere with participation in the study
* History of an autoimmune disorder or systemic inflammatory disorder
* Immunostimulatory or immunosuppressive treatment (including amphetamines or systemic corticosteroids) within 90 days
* Individuals who have ferrous metal implanted in their body other than fillings
* Individuals with current diagnoses of alcohol or substance abuse/dependence
* Anyone who is not appropriate for participation in this research protocol as deemed by the principal or co-investigator

PD Screening Questionnaire

* Do you have trouble arising from a chair?
* Is your handwriting smaller than it once was?
* Do people tell you that your voice is softer than it once was?
* Is your balance poor?
* Do your feet ever seem to get stuck to the floor?
* Do people tell you that your face seems less expressive than it once did?
* Do your arms and legs shake?
* Do you have trouble buttoning buttons?
* Do you shuffle your feet and/or take tiny steps when you walk?
* Has anyone ever told you that you have Parkinson's disease?
* Have you ever taken levodopa or Sinemet?

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 52 weeks
  An adverse event is defined as any undesirable physical, psychological, or behavioral effect experienced by a patient in conjunction with the use of the study drug.

SECONDARY OUTCOMES:
Change in UPDRS part III score | -8, -4, 0, +2, +4, +6, +8, +12 weeks
  Score from part III motor examination of the Unified Parkinson's Disease Rating Scale Score Sheet.
Change in blood analyses results | -8, -4, 0, +2, +4, +6, +8, +12 weeks
  Comprehensive metabolic panel, complete blood count with white blood cell differential (CBC/dif), and total T cell (lymphocyte) counts blood analyses
Abnormal findings in physical examination | -8, -4, 0, +2, +4, +6, +8, +12 weeks
  Physical examination including temperature, blood pressure, pulse, and skin, lung, liver, heart, and abdomen assessments.
Change in FACS results | -8, -4, 0, +2, +4, +6, +8, +12 weeks
  T cell markers analyzed by fluorescence-activated cell sorting.
Change in function of Treg cells | -8, -4, 0, +2, +4, +6, +8, +12 weeks
  Regulatory T cells isolated from peripheral blood are tested for their ability to suppress proliferation of activated T cells.
Change in magnetoencephalography (MEG) results | 0, +8, +12 weeks
  Magnetoencephalography measurements during behavioral tasks

OTHER OUTCOMES:
Change in Motion Analysis | -4, +8, +12 weeks
  Motion analysis including biomechanical assessments of the subject's mobility, postural balance, upper extremity motor control and resting state tremor.

CONTACTS AND LOCATIONS:
Overall Officials: Howard E Gendelman, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Neurology Consultants of Nebraska PC, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Background] Saunders JA, Estes KA, Kosloski LM, Allen HE, Dempsey KM, Torres-Russotto DR, Meza JL, Santamaria PM, Bertoni JM, Murman DL, Ali HH, Standaert DG, Mosley RL, Gendelman HE. CD4+ regulatory and effector/memory T cell subsets profile motor dysfunction in Parkinson's disease. J Neuroimmune Pharmacol. 2012 Dec;7(4):927-38. doi: 10.1007/s11481-012-9402-z. Epub 2012 Oct 11. PMID 23054369
- [Background] Korzenik JR, Dieckgraefe BK, Valentine JF, Hausman DF, Gilbert MJ; Sargramostim in Crohn's Disease Study Group. Sargramostim for active Crohn's disease. N Engl J Med. 2005 May 26;352(21):2193-201. doi: 10.1056/NEJMoa041109. PMID 15917384
- [Background] Reynolds AD, Stone DK, Hutter JA, Benner EJ, Mosley RL, Gendelman HE. Regulatory T cells attenuate Th17 cell-mediated nigrostriatal dopaminergic neurodegeneration in a model of Parkinson's disease. J Immunol. 2010 Mar 1;184(5):2261-71. doi: 10.4049/jimmunol.0901852. Epub 2010 Jan 29. PMID 20118279
- [Background] Mangano EN, Peters S, Litteljohn D, So R, Bethune C, Bobyn J, Clarke M, Hayley S. Granulocyte macrophage-colony stimulating factor protects against substantia nigra dopaminergic cell loss in an environmental toxin model of Parkinson's disease. Neurobiol Dis. 2011 Jul;43(1):99-112. doi: 10.1016/j.nbd.2011.02.011. Epub 2011 Mar 4. PMID 21377529
- [Background] Kim NK, Choi BH, Huang X, Snyder BJ, Bukhari S, Kong TH, Park H, Park HC, Park SR, Ha Y. Granulocyte-macrophage colony-stimulating factor promotes survival of dopaminergic neurons in the 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine-induced murine Parkinson's disease model. Eur J Neurosci. 2009 Mar;29(5):891-900. doi: 10.1111/j.1460-9568.2009.06653.x. Epub 2009 Feb 24. PMID 19245369
- [Background] McGeer PL, McGeer EG. Glial reactions in Parkinson's disease. Mov Disord. 2008 Mar 15;23(4):474-83. doi: 10.1002/mds.21751. PMID 18044695
- [Background] Benner EJ, Banerjee R, Reynolds AD, Sherman S, Pisarev VM, Tsiperson V, Nemachek C, Ciborowski P, Przedborski S, Mosley RL, Gendelman HE. Nitrated alpha-synuclein immunity accelerates degeneration of nigral dopaminergic neurons. PLoS One. 2008 Jan 2;3(1):e1376. doi: 10.1371/journal.pone.0001376. PMID 18167537
- [Background] Benner EJ, Mosley RL, Destache CJ, Lewis TB, Jackson-Lewis V, Gorantla S, Nemachek C, Green SR, Przedborski S, Gendelman HE. Therapeutic immunization protects dopaminergic neurons in a mouse model of Parkinson's disease. Proc Natl Acad Sci U S A. 2004 Jun 22;101(25):9435-40. doi: 10.1073/pnas.0400569101. Epub 2004 Jun 14. PMID 15197276
- [Background] Sheng JR, Li LC, Ganesh BB, Prabhakar BS, Meriggioli MN. Regulatory T cells induced by GM-CSF suppress ongoing experimental myasthenia gravis. Clin Immunol. 2008 Aug;128(2):172-80. doi: 10.1016/j.clim.2008.03.509. Epub 2008 May 27. PMID 18502693
- [Background] Kuhn AA, Kempf F, Brucke C, Gaynor Doyle L, Martinez-Torres I, Pogosyan A, Trottenberg T, Kupsch A, Schneider GH, Hariz MI, Vandenberghe W, Nuttin B, Brown P. High-frequency stimulation of the subthalamic nucleus suppresses oscillatory beta activity in patients with Parkinson's disease in parallel with improvement in motor performance. J Neurosci. 2008 Jun 11;28(24):6165-73. doi: 10.1523/JNEUROSCI.0282-08.2008. PMID 18550758
- [Background] Kosloski LM, Kosmacek EA, Olson KE, Mosley RL, Gendelman HE. GM-CSF induces neuroprotective and anti-inflammatory responses in 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine intoxicated mice. J Neuroimmunol. 2013 Dec 15;265(1-2):1-10. doi: 10.1016/j.jneuroim.2013.10.009. Epub 2013 Oct 29. PMID 24210793